CLINICAL TRIAL: NCT07316452
Title: Risk Prediction of Disease Progression in Early-Onset Coronary Atherosclerosis
Status: Recruiting | Type: Observational
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Principal Investigator, Zhihui Hou, Associate Director, Department of Radiology, Fu Wai Hospital, Beijing, China
Other Study IDs: 2024-2502
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Coronary Disease; Young Adult
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is part of a nationwide research project in China that aims to better understand how coronary artery disease develops and progresses in young adults. The study will enroll approximately 10,000 participants aged 45 years or younger who undergo coronary CT scans at multiple hospitals across China.

Information collected at enrollment includes basic health information, cardiovascular risk factors, blood test results, medication use, lifestyle habits, and, for some participants, genetic data. Participants will undergo follow-up coronary CT scans after several years to evaluate changes in coronary artery plaque and disease progression.

By analyzing these clinical and imaging data, the study aims to identify factors associated with disease progression and to develop prediction models that may help estimate an individual's future risk of coronary plaque progression and cardiovascular events. The results of this study may contribute to improved risk assessment and early prevention strategies for coronary artery disease in young populations.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 45 years at the time of enrollment.
2. Presence of symptoms suggestive of coronary artery disease and completion of coronary computed tomography (CT) examination.
3. Ability and willingness to provide written informed consent and to participate in follow-up assessments.

Exclusion Criteria:

1. Inability or unwillingness to complete follow-up assessments.
2. Inability to provide written informed consent.
3. History of coronary revascularization, including percutaneous coronary intervention or coronary artery bypass grafting.
4. Poor-quality coronary computed tomography images that are inadequate for reliable plaque assessment.
5. Presence of severe systemic disease with limited life expectancy that may interfere with study follow-up.
6. Pregnant or breastfeeding women.
7. Participation in another clinical study that may interfere with the outcomes of this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population includes adults aged 18 to 45 years with symptoms suggestive of coronary artery disease who undergo coronary computed tomography (CT) in participating centers across China. Participants are prospectively and consecutively enrolled into a nationwide observational registry after providing written informed consent and are followed longitudinally for disease progression.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression of Coronary Plaque on Computed Tomography | From baseline to follow-up coronary CT, up to 3 years
  Progression of coronary atherosclerotic plaque assessed by comparing baseline and follow-up coronary computed tomography scans.

CONTACTS AND LOCATIONS:
Locations (1):
- FuWai hospital, Beijing, China